CLINICAL TRIAL: NCT01129375
Title: A Randomized, Placebo-controlled, Two-period, Two-treatment, Two Sequence, Cross-over Pharmacodynamic and Pharmacokinetic Interaction Study After 5-days Repeated Oral Doses of Clopidogrel (300 mg Loading Dose Followed by 75 mg/Day) Alone or Given Concomitantly With Omeprazole 80 mg/Day in Healthy Male and Female Subjects
Brief Title: Interaction Study of Clopidogrel 300/75 mg Given Alone or Concomitantly With Omeprazole 80 mg in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: INT11146
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-12

CONDITIONS: Healthy
MeSH Terms: interventions — Clopidogrel; Omeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group clopidogrel - clopidogrel + omeprazole (Experimental): Period 1:
  * Day 1: clopidogrel 300 mg loading dose
  * Day 2 to Day 5: clopidogrel 75 mg, once daily
  Period 2:
  * Day -5 to Day -1: omeprazole 80 mg, once daily
  * Day 1: clopidogrel 300 mg loading dose + omeprazole 80 mg concomitantly
  * Day 2 to Day 5: clopidogrel 75 mg + omeprazole 80 mg concomitantly, once daily
  Each intake is under fasted conditions
  Interventions: Drug: clopidogrel; Drug: omeprazole
- Group placebo - placebo + omeprazole (Placebo Comparator): Period 1:
  * Day 1: placebo loading dose
  * Day 2 to Day 5: placebo, once daily
  Period 2:
  * Day -5 to Day -1: omeprazole 80 mg, once daily
  * Day 1: placebo loading dose + omeprazole 80 mg concomitantly
  * Day 2 to Day 5: placebo + omeprazole 80 mg concomitantly, once daily
  Each intake is under fasted conditions
  Interventions: Drug: placebo; Drug: omeprazole
- Group clopidogrel + omeprazole - clopidogrel (Experimental): Period 1:
  * Day -5 to Day -1: omeprazole 80 mg, once daily
  * Day 1: clopidogrel 300 mg loading dose + omeprazole 80 mg concomitantly
  * Day 2 to Day 5: clopidogrel 75 mg + omeprazole 80 mg concomitantly, once daily
  Period 2:
  * Day 1: clopidogrel 300 mg loading dose
  * Day 2 to Day 5: clopidogrel 75 mg, once daily
  Each intake is under fasted conditions
  Interventions: Drug: clopidogrel; Drug: omeprazole
- Group placebo + omeprazole placebo (Placebo Comparator): Period 1:
  * Day -5 to Day -1: omeprazole 80 mg, once daily
  * Day 1: placebo loading dose + omeprazole 80 mg concomitantly
  * Day 2 to Day 5: placebo + omeprazole 80 mg concomitantly, once daily
  Period 2:
  * Day 1: placebo loading dose
  * Day 2 to Day 5: placebo, once daily
  Each intake is under fasted conditions
  Interventions: Drug: placebo; Drug: omeprazole

INTERVENTIONS:
Drug: clopidogrel — Pharmaceutical form: tablet
  Route of administration: oral
  Other Names: SR25990
  Arms: Group clopidogrel + omeprazole - clopidogrel; Group clopidogrel - clopidogrel + omeprazole
Drug: placebo — Pharmaceutical form: matching tablet
  Route of administration: oral
  Arms: Group placebo + omeprazole placebo; Group placebo - placebo + omeprazole
Drug: omeprazole — Pharmaceutical form: delayed-release capsule
  Route of administration:oral

SUMMARY:
Primary objective:

* Assess the effects of clopidogrel (300 mg loading dose followed by 4 days 75 mg/day) on Adenosine diphosphate (ADP)-induced platelet aggregation when given concomitantly with omeprazole 80 mg/day compared to given alone in healthy male and female subjects

Secondary Objective:

* Compare the pharmacokinetic profiles of clopidogrel and its active metabolite when clopidogrel is given either alone or concomitantly with omeprazole

DETAILED DESCRIPTION:
The total study duration per subjects is 8 - 9 weeks broken down as follows:

* Screening: 2 to 21 days before the first dosing
* Period clopidogrel/placebo: 7 days including 5 days treatment
* Period clopidogrel/placebo + omeprazole: 12 days including 10 days treatment
* Washout between periods: at least 14 days after last dosing with respect to clopidogrel treatment
* End of study: 7 to 10 days after the last dosing

ELIGIBILITY:
Healthy subject:

* as determined by medical history, physical examination including vital signs and clinical laboratory tests:
* with a body weight between 50 kg and 95 kg if male, between 40 kg and 85 kg if female, and with a Body Mass Index (BMI) between 18 and 30 kg/m²

Exclusion Criteria:

* Evidence of inherited disorder of coagulation/hemostasis functions
* Smoking more than 5 cigarettes or equivalent per day
* Abnormal hemostasis screen
* unability to abstain from intake of any drug affecting hemostasis throughout the whole study duration
* Any contraindication to clopidogrel and/or omeprazole

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Maximum platelet aggregation intensity (MAI) induced by Adenosine diphosphate (ADP) 5µM after 5 days treatment | Day 5 of each period

SECONDARY OUTCOMES:
Maximum platelet aggregation intensity (MAI) induced by ADP 20µM after 5 days treatment | Day 5 of each period
Platelet Reactivity Index - Vasodilatator-stimulated phosphoprotein test (PRI - VASP) after 5 days treatment | Day 5 of each period
Clopidogrel pharmacokinetic parameters (maximum plasma concentration (Cmax) and area under the plasma concentration curve (AUC0-24)) after 5 days treatment | Up to 24 hours postdose on Day 5 for each period
Clopidogrel active metabolite pharmacokinetic parameters (Cmax and AUC0- 24) after 5 days treatment | Up to 24 hours postdose on Day 5 for each period

CONTACTS AND LOCATIONS:
Overall Officials: International Clinical Development Study Director, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States

REFERENCES:
- [Result] Angiolillo DJ, Gibson CM, Cheng S, Ollier C, Nicolas O, Bergougnan L, Perrin L, LaCreta FP, Hurbin F, Dubar M. Differential effects of omeprazole and pantoprazole on the pharmacodynamics and pharmacokinetics of clopidogrel in healthy subjects: randomized, placebo-controlled, crossover comparison studies. Clin Pharmacol Ther. 2011 Jan;89(1):65-74. doi: 10.1038/clpt.2010.219. Epub 2010 Sep 15. PMID 20844485